CLINICAL TRIAL: NCT00001310
Title: Immunopathology and Molecular Pathology of Ocular Diseases in Humans
Brief Title: Tissue Studies of Human Eye Diseases
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920113; 92-EI-0113
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2015-09-16

CONDITIONS: Retinal Disease; Corneal Disease; Diabetic Retinopathy; Uveitis; Age-Related Macular Degeneration
Keywords: Retinal Disease; Diabetic Retinopathy; Uveitis; Age-Related Macular Degeneration; Corneal Disease; Ocular Disease
MeSH Terms: conditions — Retinal Diseases; Corneal Diseases; Diabetic Retinopathy; Uveitis; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this project is to diagnose and evaluate ocular and related tissues with various diseases such as conjunctival, corneal, uveal, vitreoretinal and optic nerve disorders, ocular degenerative, metabolic or genetic diseases and tumors. These will be studied using light microscopy, electron microscopy, confocal microscopy, immunohistochemistry, molecular pathological including polymerase chain reaction and in situ hybridization, as well as measuring the functions of cellular organelles, e.g., mitochondrial function. Lymphocytes in the peripheral blood as well as other involved biopsied tissues and ocular tissue will be compared and categorized by disease. Cytokines, chemokines or growth factors and/or other released molecules in the blood and ocular fluids will be also analyzed. Elucidating the relationship between the infiltrating cells, ocular resident cells, and their products in various diseases will help us to make diagnoses and increase our understanding of human ocular disorders.

Patients who require eye surgery to treat an eye disease or other disease in which the eye is involved may participate in this study. Samples of eye tissue and fluid that are normally removed and discarded during eye surgery will instead be given to researchers for study. The tissues will be examined under microscope and studied using sophisticated chemical and biological tests. Immune cells from blood samples may also be examined. These studies will help better understand and diagnose the various eye diseases and to develop more attractive therapies.

DETAILED DESCRIPTION:
The purpose of this project is to diagnose and evaluate ocular and related tissues with various diseases such as conjunctival, corneal, uveal, vitreoretinal, scleral, optic nerve, and orbital disorders, ocular degenerative, inflammatory, metabolic or genetic diseases, and tumors. These will be studied using light microscopy, electron microscopy, confocal microscopy, immunohistochemistry, molecular pathology including microdissection and polymerase chain reaction and in situ hybridization, ELISA, as well as measuring the functions of cellular organelles, e.g., mitochondrial function. Lymphocytes in the peripheral blood, serum, as well as other involved biopsied tissues and ocular tissue will be compared and categorized by disease and normal. Cytokines, chemokines, growth factors, antibodies, and/or other released molecules in the blood, CSF, and ocular fluids will be also analyzed. We will compare the tissue morphology as well as immunological and biochemical indexes, e.g., cytokine/chemokine levels, growth factors, and antibodies between the diseases and normals. Elucidating the relationship between the infiltrating cells, ocular resident cells, and their products in various diseases will help us to make diagnoses, increase our understanding of human ocular disorders, and assist therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Up to 5,000 subjects will be enrolled in the study at all sites combined. Subjects will be enrolled at NEI.

1. Participants must be undergoing an eye procedure for clinical care of their condition which requires the removal of tissue specimens or have agreed pre-mortem to donate their eyes after death for research purposes.
2. Participants must agree to the de-identified storage of their sample for potential use in future research projects.
3. For conditions where blood is needed for analysis, participants must consent to having blood drawn for research evaluation, and be able to safely give a blood sample.
4. Participants must be able to give informed consent for themselves and/or their minor children who wish to enroll.

EXCLUSION CRITERIA:

1. Participant is unwilling or unable to give informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3833 (Actual)
Dates: Start 1992-03-05; Study Completion 2015-09-16

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Nussenblatt, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Chan CC. Molecular pathology of primary intraocular lymphoma. Trans Am Ophthalmol Soc. 2003;101:275-92. PMID 14971583
- [Background] Ding X, Patel M, Chan CC. Molecular pathology of age-related macular degeneration. Prog Retin Eye Res. 2009 Jan;28(1):1-18. doi: 10.1016/j.preteyeres.2008.10.001. Epub 2008 Nov 6. PMID 19026761
- [Background] Chan CC, Li Q. Immunopathology of uveitis. Br J Ophthalmol. 1998 Jan;82(1):91-6. doi: 10.1136/bjo.82.1.91. No abstract available. PMID 9536890